CLINICAL TRIAL: NCT04514575
Title: Plasma Transfusion in Major Vascular Surgery: a Danish Nationwide Registry Study
Brief Title: Plasma Transfusion in Major Vascular Surgery
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Other Study IDs: REG-144-2017
Record Dates: First submitted 2020-06-30; First posted 2020-08-17 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Aortic Aneurysm, Abdominal; Arterial Occlusive Diseases
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-FFP: Patients transfused with an FFP:RBC ratio of 2:3 to 3:3 (0.7 - 1.0)
  Interventions: Biological: Plasma transfusion
- Low-FFP: Patients transfused with an FFP:RBC ratio at or below 1:3 (0.0 - 0.3).
  Interventions: Biological: Plasma transfusion

INTERVENTIONS:
Biological: Plasma transfusion — Transfusion of allogeneic fresh frozen plasma or cryoprecipitate

SUMMARY:
BACKGROUND

* Major blood loss is frequent in open repair of ruptured and intact abdominal aortic aneurysm (AAA) as well as in aorto-bifurcated prosthesis insertion due to aortoiliac occlusive disease.
* Major blood loss is associated with death, post-operative complications and coagulopathy.
* Data from randomized trials in trauma patients indicate that a high plasma to red blood cell (RBC) transfusion ratio reduces 30-day mortality.
* No randomized trial data are available for the AAA population.
* Observational data demonstrate, that a high plasma:RBC transfusion ratio associates to a lower 30 day mortality. However, the reports are based on small cohorts of 78-165 patients, short term outcomes and lack information on major adverse events such as cardiac and respiratory.
* The Danish Vascular Registry (DVR), covering 1996-2018, contains data on approx. 4,400 ruptured and 8,200 intact (elective/symptomatic) AAA repairs, and 5,400 open aortoiliac repairs due to occlusive disease. Expected total count 1997-2018: 17,000.
* The Danish Transfusion Database (DTDB), covering approx. 1997-2018, contains information on units of RBCs, plasma and platelets transfused. A unique patient identification number (CPR) allows merging of all data set.

OBJECTIVE

To identify whether resuscitation with a high plasma to RBC ratio associates to improves survival in open abdominal aortic surgery as compared to a low plasma to RBC-ratio.

PICO

* Population: Open abdominal aortic surgery
* Intervention: "High FFP": FFP to RBC unit ratio of 2:3 to 3:3 (0.7 - 1.0)
* Comparison: "Low FFP": FFP to RBC unit ratio of 0:3 to 1:3 (0.0 - 0.3)
* Outcome: All-cause mortality 90 days following surgery.

DATA SOURCES

CPR, Danish Civil Registration System. DNPR, Danish National Patient registry. DVR, Danish Vascular registry. DPDB, The Danish national Prescription DataBase.

DETAILED DESCRIPTION:
STATISTICAL ANALYSIS PLAN

The primary analysis will be a stratified cox regression model.

STRATIFICATION:

* type of surgery/condition (ruptured AAA vs intact AAA vs aorto-iliac occlusive disease, source: DVR)
* sex (CPR)
* Center (Rigshospitalet vs. Gentofte vs. Slagelse vs. Odense vs. Kolding vs. Aarhus vs. Viborg vs. Aalborg, source: DVR)

COVARIATE ADJUSTMENT:

* calendar time (DVR)
* age (CPR)
* Carlsons comorbidity index score (DNPR)
* Priority (Acute vs. Sub-acute vs. Elective, source: DVR)
* Use of anti-thrombotic drugs (DPDB). A covariate of 4 levels (ATC code is noted in parenthesis).

  1. None vs.
  2. Anti-platelet therapy

     * acetylsalicylic acid (B01AC06) or
     * dipyridamole (B01AC07, eg. persantin or asasantin)
  3. Anti-platelet therapy "thienopyridines-like drugs"

     * clopidogrel (B01AC04) or
     * ticagrelor (B01AC24, eg. Brilique) or
     * prasugrel (B01AC22, eg. Efient) Comment: patients prescribed thienopyridines in combination with aspirin will be included in this "thienopyridine anti-platelet group 3"
  4. Anti-coagulant therapy

     * Vitamin K antagonists (B01AA, eg. warfarin or phenprocoumon)
     * Low-molecular weight heparine (B01AB01-10)
     * Direct thrombin inhibitors (B01AE, eg. Pradaxa/Dabigatran)
     * Direct factor Xa inhibitors (B01AF, eg. Rivaroxaban/Xarelto). Comment: patients prescribed both anticoagulant- and antiplatelet therapy and will be included in this "Anti-coagulant group 4".

ADDITIONAL ANALYSES:

1. Stratify the population into 4 groups according to the total transfusion requirement

   1. patients receiving 10 units or less of any blood product < 24 hrs or 11-15 units < 48 hrs.vs.
   2. patients receiving 11-15 units of any blood product < 24 hrs. or 16-20 units < 48 hrs. vs.
   3. patients receiving 16-20 units of any blood product < 24 hrs. or 21-25 units < 48 hrs. vs.
   4. patients receiving more than 20 units of any blood product < 24 hrs. or more than 25 units < 48 hrs.
2. Outcome predicted by a joint function (general interaction) of total plasma transfusion and total blood cell transfusion will be assessed in an exploratory way by inspection and by agnostic modelling in the mold of Multivariate Adaptive Regression Splines (MARS) and recursive partitioning, i.e. Classification And Regression Trees (CART).
3. Redefine intervention and control group as 4th and 1st quartile of FFP:RBC ratio. Initially, the population will be divide into 4 groups according to quartiles and compared the population below 1st quartile with the population above the 4th quartile, which will define the low vs. the high FFP group, resp. However, to allow for stratification for operation type (ruptured AAA vs. intact AAA vs. occlusive disease) it may be necessary to adjust the percentile cut to retain power in the analyses. For instance, the population may be cut according to tertiles, or, if there is sufficient data, cut by quintiles (5 groups) or deciles (10 groups).
4. Confine the population to patient with blood loss above 50 % of total blood volume (calculated by Naddler's equation accounting for sex, weight and height). If height and weight are not available, the registered blood loss must exceed 2 L in females and 2.5 L in males.
5. Adjusting exclusively for calendar year, sex, age, Charlson's comorbidity index score, and center (ie, excluding priority and antithrombotic therapy).

MISSING DATA

Missing data will not be an issue for the number of blood transfusions because units of blood products transfused are used as an inclusion criterion. All remaining covariates are discrete, and missing data for each of those will be included as separate parameters (factor level).

STATISTICAL SIGNIFICANCE LEVEL

Bonferroni adjustment of the significance level will be applied to control for multiple testing.

With one primary and four secondary outcomes, only a P-value below 0.01 (0.05/5) will be considered statistically significant. A P-value between 0.01 and 0.05 will be considered borderline significant.

ELIGIBILITY:
Inclusion Criteria:

1. Open abdominal aortic repair with the insertion of prosthesis for either

   * intact (elective or symptomatic) AAA
   * ruptured AAA
   * aorto-iliac occlusive disease
2. Requiring massive transfusion defined as 10 units or more of any blood product(*) transfused on the same date (source DTDB)

(*) = Allogeneic packed RBCs, FFP, cryoprecipitate, or platelets. Cryoprecipitate will account for 4 units of FFP in the FFP:RBC ratio.

Exclusion Criteria:

1. Surgery time limited to < 50 minutes (DVR)
2. No prosthesis inserted (DVR) AND operation date (DVR) equal to the death date (CPR)

Excluding patients with surgery time less than 50 minutes or cases where no prosthesis has been inserted is expected to minimize survival bias from patients exsanguinating in the operation theater before blood products can be delivered. Intentionally, it may also exclude cases where surgery was considered futile and halted.

Ages: 41 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Denmark, every citizen is registered with a unique identification number in the Civil Registration System. Patients undergoing major open abdominal aortic surgery (above 40 and below 100 years of age) registered in the Danish Vascular Registry in the period between January 1st 1997 and December 31st 2018 will be identified and linked to national health registers by using the unique identification number. The DTDB will provide data on blood transfusions. The DNPR will provide data on complications by ICD10 code and on hospital admission duration.
  Data sources CPR, Danish Civil Registration System. DNPR, Danish National Patient registry. DVR, Danish Vascular registry. DPDB, The Danish national Prescription DataBase.
Sampling Method: Probability Sample
Enrollment: 17000 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
90-day survival | First 90 days after index surgery
  Survival data. Source: CPR

SECONDARY OUTCOMES:
30-day survival | First 30 days after index surgery
  Survival data. Source: CPR
1-year survival | 1 year after index surgery
  Survival data. Source: CPR
Death or any major adverse events at 90-days | First 90 days after index surgery
  Dichotomous outcome. Source: DNPR and DVR.
  A. Major adverse cardiovascular events "MACE" [ICD10-codes]
  * acute myocardial infarction [DI21.0-23.9, DT817Y2]
  * stroke [DI60-64.9, DT817Y1]
  * non-fatal cardiac arrest [DI460]
  B. Major adverse respiratory events
  * adult respiratory distress syndrome [DJ80]
  * pulmonary edema [DJ81]
  * pulmonary embolism [DI26, DT817D]
  C. Major adverse vascular event
  * bowel ischemia [DK550C-H]
  * vascular reoperation for deep rebleeding or thrombus or embolus [KPWE, KPWG], lower-limb fasciotomy [KNGM09, KNHM09, KNFM09] or explorative laparotomy [KJAH00]
  * major lower limb amputation [KNE-HQ]
  * acute limb ischemia requiring intervention
  D. Other
  * renal replacement therapy [BJFD, DZ992]
  * AB0-incompatibility reaction [DT803]
  * Rhesus-incompatibility reaction [DT804]
  * Hemorrhage and hematoma complicating a procedure, not elsewhere classified [T810, DT810G, DT810E]
Number of days alive outside hospital within 90 days | Day 90 after index surgery
  Count data. Source: DNPR and CPR

CONTACTS AND LOCATIONS:
Overall Officials: Ole Pedersen, MD, PhD, Study Director — Department of Clinical Immunology, Naestved Hospital, Denmark.
Locations (1):
- Slagelse Hospital, Slagelse, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desborough M, Sandu R, Brunskill SJ, Doree C, Trivella M, Montedori A, Abraha I, Stanworth S. Fresh frozen plasma for cardiovascular surgery. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD007614. doi: 10.1002/14651858.CD007614.pub2. PMID 26171897
- [Background] Holcomb JB, Tilley BC, Baraniuk S, Fox EE, Wade CE, Podbielski JM, del Junco DJ, Brasel KJ, Bulger EM, Callcut RA, Cohen MJ, Cotton BA, Fabian TC, Inaba K, Kerby JD, Muskat P, O'Keeffe T, Rizoli S, Robinson BR, Scalea TM, Schreiber MA, Stein DM, Weinberg JA, Callum JL, Hess JR, Matijevic N, Miller CN, Pittet JF, Hoyt DB, Pearson GD, Leroux B, van Belle G; PROPPR Study Group. Transfusion of plasma, platelets, and red blood cells in a 1:1:1 vs a 1:1:2 ratio and mortality in patients with severe trauma: the PROPPR randomized clinical trial. JAMA. 2015 Feb 3;313(5):471-82. doi: 10.1001/jama.2015.12. PMID 25647203
- [Background] Johansson PI, Stensballe J, Rosenberg I, Hilslov TL, Jorgensen L, Secher NH. Proactive administration of platelets and plasma for patients with a ruptured abdominal aortic aneurysm: evaluating a change in transfusion practice. Transfusion. 2007 Apr;47(4):593-8. doi: 10.1111/j.1537-2995.2007.01160.x. PMID 17381616
- [Background] Mell MW, O'Neil AS, Callcut RA, Acher CW, Hoch JR, Tefera G, Turnipseed WD. Effect of early plasma transfusion on mortality in patients with ruptured abdominal aortic aneurysm. Surgery. 2010 Nov;148(5):955-62. doi: 10.1016/j.surg.2010.02.002. Epub 2010 Apr 7. PMID 20378142
- [Background] Mesar T, Larentzakis A, Dzik W, Chang Y, Velmahos G, Yeh DD. Association Between Ratio of Fresh Frozen Plasma to Red Blood Cells During Massive Transfusion and Survival Among Patients Without Traumatic Injury. JAMA Surg. 2017 Jun 1;152(6):574-580. doi: 10.1001/jamasurg.2017.0098. PMID 28273299
- [Background] Montan C, Hammar U, Wikman A, Berlin E, Malmstedt J, Holst J, Wahlgren CM. Massive Blood Transfusion in Patients with Ruptured Abdominal Aortic Aneurysm. Eur J Vasc Endovasc Surg. 2016 Nov;52(5):597-603. doi: 10.1016/j.ejvs.2016.07.023. Epub 2016 Sep 4. PMID 27605360
- [Background] Sperry JL, Guyette FX, Adams PW. Prehospital Plasma during Air Medical Transport in Trauma Patients. N Engl J Med. 2018 Nov 1;379(18):1783. doi: 10.1056/NEJMc1811315. No abstract available. PMID 30380388

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04514575/Prot_SAP_001.pdf